CLINICAL TRIAL: NCT02631486
Title: Does Early Mobilisation After Surgical Repair of Rotator Cuff Tears Improve Biomechanical and Clinical Outcomes?
Brief Title: Does Early Mobilisation Improve Outcomes After Rotator Cuff Repair?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Lancashire (Other)
Collaborators: Wrightington, Wigan and Leigh NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Bruno Fles Mazuquin, Mr, University of Central Lancashire
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STEMH 277
Record Dates: First submitted 2015-12-10; First posted 2015-12-16 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Shoulder; Rehabilitation
Keywords: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early (Experimental): The first group will use sling for comfort only. Active assisted exercises in closed chain and in safe zone are allowed in the first 4 weeks.
  The rehabilitation stages will start from active assisted progressing to more active stages phases until full recovery. The whole program will last about 3 months.
  Interventions: Other: Physiotherapy
- Conservative (Active Comparator): The second group will use a sling for 6 weeks. The rehabilitation stages will start with active assisted/closed chain movements with short levers, it will progress to more active stages phases until full recovery. The whole program will last about 3 months.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Passive exercises, active exercises, strengthening, stretching

SUMMARY:
Shoulder pain is among the most common musculoskeletal complaints, leading to high number of General Practioners consultations in the United Kingdom. On the top list of the disorders causing pain and dysfunction of shoulder is rotator cuff tears. The aetiology of rotator cuff tears is multifactorial and is likely to be a combination of age-related degenerative changes and trauma during life. It is present in approximately 25% of individuals in their 60s and 50% of individuals in their 80s and have been shown to start developing during the 40s. To recover functional status of this patients group, surgical repair is often recommended, but for optimal results the rehabilitation is of great importance and must be adequately planned. After surgery a period of movement restriction is followed, however, the optimal time of immobilisation is unknown. As a common practice, patients use a sling for six weeks and avoid any activities with the affected shoulder. This period is important to protect the tendon, allow good healing and to possibly prevent re-tear episodes. Although, the delayed motion may increase the risk of postoperative shoulder stiffness, muscle atrophy and potentially delay improvement of functionality. Based on the available evidence, it is difficult to make a clinical decision for a well-programmed rehabilitation regime and establish the most favourable postoperative time to start it. Moreover, it is not clear if early mobilisation will benefit more severe stages as published studies have methodological flaws that compromises the clinical decision for patients with higher commitments. The question whether early mobilisation application is beneficial is of high importance as the results will not just help improving patients quality of life, but also may reduce costs as further complication may be avoided.

DETAILED DESCRIPTION:
The study will be a randomised controlled trial, which means that each participant will have equal chances to be assigned to one of 2 groups.

The first group will start the rehabilitation after 3 weeks post-surgery and the second group will start after 6 weeks.

The rehabilitation stages will start with passive movements, progressing to more active stages phases until full recovery. The whole program will last about 3 months, which is in accordance to what is normally used at the Wrightington Hospital.

Each participant will have 4 assessment sessions: 1 pre-surgery, after 3 months post-surgery, after 6 months and the last after 12 months post-surgery.

The assessment sessions will consist on answering questionnaires and a clinical assessment with equipment, which measures muscle activity and joint angles during clinical tasks.

An ultrasound scan of the shoulder to assess the integrity of the rotator cuff would be carried out one year after surgery by a consultant radiologist.

These assessments are timed with the routine orthopaedic clinic assessments so that patients do not have to make extra trips to take part in the research.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 70 years old,
* Confirmed diagnosis of rotator cuff tear
* No previous shoulder surgery
* No other musculoskeletal impairment in the assessed limb or cervical and thoracic spine.

Exclusion Criteria:

* Previous shoulder surgery
* Fixation which does not allow early mobilisation
* Other musculoskeletal impairment in the assessed limb or cervical and thoracic spine,
* People with special needs who are unable to understand the instructions needed,
* Non-English or non-Portuguese speakers.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04; Primary Completion 2018-04 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline range of motion | Pre-surgery (baseline), change from baseline range of motion at 3 months, change from baseline range of motion at 6 months, change from baseline range of motion at 1 year

SECONDARY OUTCOMES:
Change from baseline muscle activity in millivolts | Pre-surgery (baseline), change from baseline range of motion at 3 months, change from baseline range of motion at 6 months, change from baseline range of motion at 1 year
  The muscle activity will be measured using non-invasive electromyography
Re-tears ratio | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jim Richards, Professor, Principal Investigator — University of Central Lancashire
Locations (1):
- Wrightington Hospital, Wigan, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No